CLINICAL TRIAL: NCT00265954
Title: A Randomized Trial of an Internet Versus In-person Behavioral Weight Loss Treatment Program.
Brief Title: Internet Assisted Obesity Treatment
Acronym: iReach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Arkansas (Other)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Interim Dean, College of Agriculture and Life Sciences, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK56746; R01DK056746 (NIH)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

ARMS (3):
- 1 (Experimental): Individuals in this arm receive a 6 month behavioral weight loss intervention delivered on-line. Groups meet via a web chat weekly for 24 weeks and monthly for the following 12 months.
  Interventions: Behavioral: internet, in-person and internet+in-person
- 2 (Experimental): In-person; Individuals in the in-person condition attend weekly group behavioral weight loss sessions for 24 weeks and then monthly sessions for the following 12 months.
  Interventions: Behavioral: internet, in-person and internet+in-person
- 3 (Experimental): In-person+internet; Individuals in this condition receive a behavioral weight loss intervention over the internet weekly for 24 weeks and monthly for the following 12 months. Every month during the first 24 weeks and every third month during the following year they have an in-person meeting.
  Interventions: Behavioral: internet, in-person and internet+in-person

INTERVENTIONS:
Behavioral: internet, in-person and internet+in-person — All participants receive an 18 month behavioral weight loss program that meets weekly for the first 6 months and monthly for the next year.

SUMMARY:
High quality behavioral weight loss programs are not widely accessible. The Internet offers one way to deliver health behavior programs to a wider audience. However, effective weight loss treatments are intensive and program delivery over the Internet may not be capable of duplicating the level of engagement typically generated during traditional in-person treatment. The goal of this study is to test the effectiveness of three weight loss interventions: Internet alone, Internet+periodic in-person support, and in-person alone. The investigators hypothesize that the in-person and internet+in-person interventions will produce better weight loss and maintenance than the internet only group.

DETAILED DESCRIPTION:
Currently 65% of the adult population is overweight or obese. Unfortunately, safe and effective treatments for obesity are costly and intensive; therefore, this level of support is unlikely to be feasible in most clinical settings. Moreover, an additional limitation to current obesity treatment approaches is the limited reach and availability of programs for persons who work, live in rural areas or do not want, or cannot afford participation in group support classes. The advent of telecommunications technology may provide a solution to this dilemma. Telecommunications technology can presumably improve access to services and improve efficiency of delivery. Moreover, research examining new technologies such as the Internet, will provide information for policy makers interested in disseminating low-cost, high reach effective obesity treatment interventions. However, the effectiveness of the Internet for inducing weight loss has not been rigorously tested. Therefore, the overall goal of this project is to determine if obesity treatment can be effectively delivered over the Internet. A secondary aim is to evaluate whether the effectiveness of Internet interventions can be improved with the addition of minimal in-person support. Specifically, this project is a randomized, controlled clinical trial designed to test the translation of a behavioral weight loss program to the Internet (I). The I intervention will be compared to both an in-person condition (IP) and an Internet condition supplemented with periodic in-person support (I+IP). Subjects will be 488 (30% minority) overweight and obese adults recruited from Vermont and Arkansas who will participate in a 6-month behavioral weight control treatment program followed by 12 months of weight maintenance. Assessments will include measures of body weight, adherence to treatment goals, social influence components and frequency of use of Internet website features.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* BMI>25
* Internet access

Exclusion Criteria:

* pregnancy
* major medical problems
* inability to walk for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2006-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Body Mass Index or body weight change | 0, 6, 12, 18 month time points

SECONDARY OUTCOMES:
Social support, diet, exercise, adherence to treatment components | 0, 6, 12, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Harvey-Berino, PhD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - University of Arkansas for the Medical Sciences, Little Rock, Arkansas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Harvey-Berino J, Krukowski RA, Buzzell P, Ogden D, Skelly J, West DS. The accuracy of weight reported in a web-based obesity treatment program. Telemed J E Health. 2011 Nov;17(9):696-9. doi: 10.1089/tmj.2011.0032. Epub 2011 Sep 1. PMID 21882997